CLINICAL TRIAL: NCT01528878
Title: A Dose-finding, Safety and Preliminary Efficacy Study of Stereotactic Radiosurgery for Hepato-cellular Carcinoma and Metastatic Disease to the Liver.
Brief Title: Safety, Efficacy, and Dosing of Stereotactic Radiosurgery for Hepato-cellular Carc/Colo-rectal Liver Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0809
Record Dates: First submitted 2012-01-09; First posted 2012-02-08 (Estimated); Results first posted 2018-05-15 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Liver Neoplasms; Colonic Neoplasms; Metastatic Cancer to Liver
Keywords: Liver Cancer; Hepatocellular Carcinoma; HCC; Metastatic Cancer to Liver; Metastatic Colon Cancer; Metastatic Colo-rectal Cancer; mCRC; Liver Function; Child-Pugh
MeSH Terms: conditions — Liver Neoplasms; Colonic Neoplasms; Carcinoma, Hepatocellular | interventions — Radiotherapy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Good liver function. (Experimental): Patients with good liver function as defined by no more than Child-Pugh Class A.
  Interventions: Radiation: Stereotactic Radiosurgery using the CyberKnife System.
- Compromised liver function. (Experimental): Patients with compromised liver function as defined by patients with Child-Pugh Class B.
  Interventions: Radiation: Stereotactic Radiosurgery using the CyberKnife System.

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery using the CyberKnife System. — Radiation: Stereotactic Radiosurgery using the CyberKnife System. The CyberKnife system has been cleared by the U.S. Food and Drug Administration (FDA) to treat lesions, tumors and conditions, anywhere in the body when radiation treatment is indicated. To address movement of target lesion during the respiratory cycle, the Synchrony™ option will be used.
  The Synchrony option precisely tracks tumors in or near the target organ as they move, enabling the highly focused beams of radiation to destroy the tumors with minimal injury to adjacent normal tissue. The Synchrony option records the breathing movements of a patient's chest and combines that information with sequential x-ray pictures of tiny markers inserted inside or in the proximity of the tumor to enable precise delivery of radiation during any point in the respiration cycle. The CyberKnife system with the Synchrony option enables reduced normal tissue exposure by using smaller treatment margins and increased accuracy.
  Other Names: Radiotherapy; CyberKnife; Stereotactic Radiosurgery

SUMMARY:
The purpose of this study is to determine a tolerable dose of radiation delivered by the CyberKnife system in two groups of patients with hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
The CyberKnife system has been cleared by the U.S. Food and Drug Administration (FDA) to treat lesions, tumors and conditions anywhere in the body when radiation treatment is indicated. In order to treat tumors during the respiratory cycle (vs. increasing the margin of treatment around the tumor to compensate for movement or requiring the patient to breath hold during the delivery of each beam), the Synchrony™ option, a system option that enables dynamic radiosurgery during respiration, will be used. The purpose of this study is to determine a tolerable dose of radiation delivered by the CyberKnife in two groups of patients with hepatocellular carcinoma (HCC).Group 1: Patients with HCC and Childs A cirrhosis, and patients with colorectal liver metastases. Group 2: Patients with Childs B cirrhosis. Patients will be irradiated with radiation doses using the CyberKnife system in 3-5 radiation fractions using guidance from fiducials placed by interventional radiology. Treatments will be delivered with standard CyberKnife procedures to account for respiratory motion and set up variations. The fiducial location will be the prime determinant of the delivery site and respiratory motion and fiducial markers will be placed via percutaneous approach by interventional radiology.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatocellular carcinoma (as defined by biopsy or alpha-fetoprotein (AFP) greater than 1000ng/dL with appropriate imaging) or liver metastases from colorectal cancer or other tumor (as defined by biopsy or elevated Carcinoembryonic antigen (CEA) or a positive positron emission tomography (PET) scan in conjunction with a mass on CT or MRI in a patient with previously resected cancer). Patients with at least one measurable liver lesion and no more than 3 are eligible if they meet all other eligibility criteria including the dose constraints on the composite plan.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
3. Patients are not candidates for definitive surgical resection because of tumor location, hepatic function, or other medical or personal reasons.
4. Patients with HCC who are being considered for liver transplant may be entered as a bridge to transplant if it is considered by the transplant team that an ablative therapy would be of value while awaiting transplant.
5. If cirrhosis is present, patients will have Child-Pugh score of A or B (see Appendix A in the Master Protocol).
6. Patients will have tumors not optimally treated with radio-frequency ablation by interventional radiology, or by GI/transplant surgery. This could be for reasons of size, tumor location, or other reasons.
7. Ability to place fiducial markers in the vicinity of the tumor to allow for radiographic tracking of respiratory motion and tumor localization. Fiducial placement will generally be done by interventional radiology.
8. Estimates of hepatic tolerance must meet the criteria as defined in Section III. This eligibility will not be able to made definitively until the patient has agreed to participate. in the study and the appropriate scan analyses and dosimetry have been performed. No more than one decrement in dose from the planned dose level will be allowed for an individual patient because of exceeding the maximal liver doses before the patient is declared ineligible for study.
9. Adequate bone marrow and renal function as assessed by the following:

   * Absolute neutrophil count (ANC) > 1000/mm3
   * Platelet count > 80,000/mm3
   * Creatinine < 2.0 mg/dL OR Creatinine clearance > 45 mL/min based on Cockcroft-Gault formula).
10. Patients with extra hepatic metastatic disease are eligible if it is the opinion of the treating physician that local therapy to the liver may produce worthwhile clinical benefits
11. Patient is able to understand fully the potential risks and benefits of this approach and signs an appropriate informed consent.
12. Male and female of >18 years of age. Male or female patients capable of reproduction must agree to use medically acceptable methods of contraception, such as an intrauterine device, diaphragm, with spermicide, condom with spermicide or abstinence. Inclusion of females of childbearing potential requires a negative pregnancy test within 14 days prior to study initiation.

Exclusion Criteria:

1. Child-Pugh Class C cirrhosis
2. Patients with clinically apparent central nervous system (CNS) disease.
3. Medical or psychiatric illness that would not allow the patient to tolerate the proposed treatment including inability to lie flat for an extended period of time, severe claustrophobia or other reasons.
4. Uncontrolled or significant cardiovascular disease including: myocardial infarction within 6 months, uncontrolled angina within 6 months, Class III-IV New York Heart Association (NYHA) congestive heart failure, grade 3 cardiac valve dysfunction
5. Evidence of decompensated liver disease as evidenced by: clinically significant ascites refractory to diuretic therapy) evidence of hepatic encephalopathy, coagulopathy not corrected by conservative measures.
6. A history of CTCAE Grade 3 bleeding esophageal or gastric varices within the past 2 months. Prior variceal bleed permitted if patient has undergone banding or sclerotherapy and there has been no evidence of bleeding for 2 months. Patients at risk for varices (based on the following: known history of esophageal or gastric varices; evidence of hepatic cirrhosis and/or portal hypertension including biopsy-proven cirrhosis, hypersplenism, or radiographic findings of varices) will be screened for esophageal varices. If varices are identified that require intervention (banding), patient will not be eligible until varices adequately treated.
7. Prisoners or patients who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.
8. Uncontrolled intercurrent illness.
9. Inability to comply with study and/or follow-up procedures.
10. A patient with Child-Pugh Class A will not be eligible for study if the liver dose constraint described in Section 3.2 cannot be met after two decrements in dose per fraction as described above.
11. A patient with Child-Pugh Class B will not be eligible for study if the liver dose constraint described in Section 3.2 cannot be met after two decrements in dose per fraction as described above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2014-08-18 (Actual); Study Completion 2016-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Tepper, MD, Principal Investigator — University of North Carolina at Chapel Hill Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - East Carolina Medical School, Greenville, North Carolina

REFERENCES:
- See also: Website for University of North Carolina Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from June, 2009 to March, 2014 at two institutions.
Pre-assignment Details: 39 participants were consented and 9 were found ineligible and were not treated.
Groups:
- Single Arm Patients With HCC or Liver Metastases: Patients with hepatocellular carcinoma (HCC) who are not appropriate for surgical resection or radiofrequency ablation (RFA) as a bridge to transplant. The original cohort was not analyzed between good vs compromised liver function because there were only 2 patients with Child-Pugh Class B and secondary outcomes measured are thought to be more influenced by disease rather than liver function (which may be more relevant for toxicity).
Period: Overall Study
Arm/Group | Single Arm Patients With HCC or Liver Metastases
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The original cohort was not analyzed between good vs compromised liver function because there were only 2 patients with Child-Pugh Class B and secondary outcomes measured are thought to be more influenced by disease rather than liver function (which may be more relevant for toxicity).
Arm/Group | Single Arm Patients With HCC or Liver Metastases
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 65.5 [23 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Measure Description: A scale from 0-5 to describe a patient's level of functioning in terms of selfcare ability and activity level.
  0, Fully active
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 17
    1 | 13
Child Pugh Score [Count of Participants; unit: Participants] — The Child-Pugh score consists of five clinical features and is used to assess the prognosis of chronic liver disease and cirrhosis. The score employs five clinical measures of liver disease. Each measure is scored 1-3, with 3 indicating most severe derangement.
  Child- Pugh Class:
  A 5-6 points B 7-9 points C >9 points
  Participants
    5 (Class A) | 22
    6 (Class A) | 6
    >=7 (Class B) | 2
Primary Disease [Count of Participants; unit: Participants]
  Hepatocellular carcinoma | 11
  Metastatic cancer | 19
Prior liver-directed therapies [Count of Participants; unit: Participants]
  Any local therapy | 14
  Liver resection | 9
  Trans-arterial chemoembolization (TACE) | 7
  Radiofrequency ablation (RFA) | 6
  > 1 prior local therapy | 9
  Resection + RFA | 3
  Resection + TACE | 2
  Resection x2 + RFA | 1
  TACE + RFA x3 | 1
  TACE x 2 + RFA | 1
  TACE x 2 | 1
Prior systemic therapy [Count of Participants; unit: Participants] | 16
Number of lesions treated [Count of Participants; unit: Participants]
  1 | 26
  2 | 3
  3 | 1
Lesion size (cm) [Count of Participants; unit: Participants]
  <2 | 1
  2-2.9 | 10
  3-3.9 | 9
  4-4.9 | 2
  5-5.9 | 5
  >6 | 3
Lesion size (cm) median (range) [Median (Full Range); unit: cm] | 3.5 [1.7 to 6.5]
Gross tumor volume (cc) median (range) [Median (Full Range); unit: cc] — The demonstrable extent of a tumor seen or felt with standard examination techniques. The gross tumor volume is used in radiation oncology as the basis for initial estimates of the extent of a tumor that will undergo treatment with external beam radiation or brachytherapy
  cc | 22.5 [2.8 to 145]
Planning target volume (cc) median (range) [Median (Full Range); unit: cc] — Planning target volume (PTV) is created by expanding gross tumor volume (GTV) by 0.5-0.8 cm in all directions
  cc | 65.5 [17.7 to 258.1]
Fractionation [Count of Participants; unit: Participants] — When the total dose of radiation is divided into several, smaller doses over a period of several days, there are fewer toxic effects on healthy cells
  Participants
    5.5 Gy x 5 = 27.5 Gy | 1
    7 Gy x 5 = 35 Gy | 2
    10 Gy x 3 = 30 Gy | 1
    12.5 Gy x 3 = 37.5 Gy | 4
    13.33 Gy x 3 = 40 Gy | 1
    15 Gy x 3 = 45 Gy | 21
Dose of Radiation Therapy (Gy) [Median (Full Range); unit: Gray (Gy)] | 45 [27.5 to 45]
Mean liver dose (Gy) ) [Median (Full Range); unit: Gy] | 10.3 [4.4 to 16.5]
Volume of liver receiving <15 Gy (cc) [Median (Full Range); unit: cc] | 1239 [721 to 2289]

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Stereotactic Body Radiotherapy (SBRT) Based on Number of Cumulative Acute Toxicities Occurring Within 90 Days of Treatment and Related to SBRT.
Description: To determine a tolerable dose, cumulative acute toxicity was collected (defined as toxicity occurring within 90 days of treatment initiation). Adverse events were graded by the Common Terminology Criteria for Adverse Events version 3.0. Tolerability was based on hepatic toxicity. A grading (severity) scale is provided for each adverse event (AE) term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Groups:
- Grade 2 Adverse Events: Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL)
- Grade 3 Adverse Events: Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
Arm/Group | Grade 2 Adverse Events | Grade 3 Adverse Events
Number analyzed (Participants) | 30 | 30
Participants
  Elevated Aspartate Aminotransferase | 5 | 1
  Elevated Bilirubin | 4 | 0
  Low Hemoglobin | 4 | 0
  Fatigue | 4 | 0
  Increased Alanine Aminotransferase | 3 | 0
  Decreased Leukocyte | 2 | 1
  Nausea | 2 | 0
  Abdominal pain | 2 | 0
  Increased alkaline phosphatase | 2 | 0
  international normalized ratio increased | 2 | 0
  Decreased Platelets | 2 | 0
  Dyspnea | 1 | 0
  Acute total | 14 | 2

2. Secondary Outcome: Local Tumor Control to Doses of Radiation in Patients With Liver Cancer or Metastases to the Liver
Description: 1 year local control defined as percentage of patients with freedom from local progression at a median follow-up time of 12.7 months. Progressive disease is defined as increase by >= 50% of product of the two perpendicular diameters of an irradiated lesion.
Time Frame: 12.7 months
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm Patients With HCC or Liver Metastases
Number analyzed (Participants) | 30
percentage of participants | 81

3. Secondary Outcome: Percentage of Local Response to Doses of Radiation in Patients With Liver Cancer or Metastases to the Liver
Description: Complete response (CR) is defined as disappearance of the target lesion, partial response (PR) as regression of measureable disease, progressive disease (PD) as increase by >= 50% in product of the two perpendicular diameters of an irradiated lesion, and stable disease (SD) as all others not meeting criteria for CR, PR, or PD.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm Patients With HCC or Liver Metastases
Number analyzed (Participants) | 30
percentage of participants
  Complete Response | 7
  Partial Response | 13
  Stable Disease | 80

4. Secondary Outcome: Overall Survival of Patients With Liver Cancer or Metastases to the Liver
Description: Overall survival is defined as percentage of patients remaining alive from start of study treatment to 1 year.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm Patients With HCC or Liver Metastases
Number analyzed (Participants) | 30
percentage of participants | 62

ADVERSE EVENTS:
Time Frame: 44 weeks
Arm/Group | Single Arm Patients With HCC or Liver Metastases
All-Cause Mortality (participants affected / at risk) | 15/30
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Patients With HCC or Liver Metastases (N=30)
Pain- chest wall (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Patients With HCC or Liver Metastases (N=30)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 7
Alkaline phosphatase (Investigations) | 13
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 9
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 14
Bilirubin (hyperbilirubinemia) (Investigations) | 7
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Edema: limb (General disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 16
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4
Hemoglobin (Blood and lymphatic system disorders) | 7
INR (International Normalized Ratio of prothrombin time) (Investigations) | 3
Leukocytes (total WBC) (Investigations) | 7
Lymphopenia (Investigations) | 14
Mood alteration - Anxiety (Psychiatric disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4
Pain - Abdomen NOS (Gastrointestinal disorders) | 7
Pain - Back (Musculoskeletal and connective tissue disorders) | 4
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 3
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 2
Platelets (Investigations) | 11
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-12-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT01528878/Prot_SAP_000.pdf